CLINICAL TRIAL: NCT02794467
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind, Parallel Group, Proof of Concept Study With an Interim Futility Analysis of Epelsiban in Patients With Adenomyosis
Brief Title: Placebo-controlled Proof of Concept Study of Epelsiban in Women With Adenomyosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was prematurely discontinued due to GSK's change in prioritization for the portfolio and is not due to any safety concerns or regulatory interaction.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201580
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Adenomyosis
Keywords: Heavy menstrual bleeding; Adenomyosis; Safety; Epelsiban; Tolerability; Proof of concept
MeSH Terms: conditions — Adenomyosis; Menorrhagia | interventions — epelsiban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epelsiban 75 mg (Experimental): Approximately 24 subjects will receive 75 mg of epelsiban three times a day (TID) via oral administration
  Interventions: Drug: Epelsiban
- Epelsiban 200 mg (Experimental): Approximately 24 subjects will receive 200 mg of epelsiban TID via oral administration
  Interventions: Drug: Epelsiban
- Placebo (Placebo Comparator): Approximately 24 subjects will receive a matching placebo TID via oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epelsiban — Epelsiban will be supplied as modified capsule shaped, white coated, oral tablet with a unit dose strength of 25 or 150 mg; to be taken with food or immediately after a meal, without chewing
  Arms: Epelsiban 200 mg; Epelsiban 75 mg
Drug: Placebo — A matching placebo will be supplied as modified capsule shaped, white coated, oral tablet; to be taken with food or immediately after a meal, without chewing.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the efficacy, safety, and tolerability of epelsiban compared with placebo in treatment of women with adenomyosis.

This is a 12-week, randomized, double-blind, placebo-controlled, parallel group study with an interim futility analysis. Subjects will be randomized 1:1:1 to receive 75 milligrams (mg) of epelsiban three times daily (TID), 200 mg of epelsiban TID, or placebo TID. The study will be composed of three periods: screening, treatment, and follow-up and the total time a subject will be in the study will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen to 55 years of age, inclusive
* Pre-menopausal with a history of regular menstrual cycles every 21-35 days and without intermenstrual bleeding heavier than spotting and staining.
* Females with adenomyosis confirmed on magnetic resonance imaging (MRI), - Females with heavy menstrual bleeding .
* Willing and able to collect all menstrual cycle by-products for each cycle from screening to follow up.
* Not pregnant as confirmed by a negative serum human chorionic gonadotropin

Exclusion Criteria:

* A female subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Abnormal gynecological examination other than adenomyosis and/or breast examination requiring intervention within six months of study start
* Abnormal endometrial biopsy within six months of starting study treatment.
* History of an endometrial ablation within 12 months of starting study treatment.
* Uterine artery embolization within six months of starting study treatment.
* Prior major uterine procedures or any other significant uterine abnormalities on MRI (previous caesarean section, dilation and curettage, and diagnostic hysteroscopy are permitted).
* Confirmed rectovaginal endometriosis in women who have undergone a prior laparoscopy.
* Active pelvic infection or current use of an intrauterine device within three months of screening.
* Women with a history of transfusion for heavy menstrual bleeding within the past 2 years or history of postpartum hemorrhage.
* Any uterine dimension >20 centimeter (cm).
* Other major causes of heavy menstrual bleeding -
* Use within 3 months or anticipated use of medications that modify reproductive function
* Use or anticipated use of the following drugs: anticoagulants aminocaproic acid ,or any other medications that affect menstrual bleeding such as tranexamic acid.
* Use of daily opioid pain medications other than with menses.
* Hemoglobin <8 grams (g)/deciliter.
* History of bleeding disorder or known presence of acquired or inherited thrombophilia, (sickle cell trait individuals are not excluded).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Mean percent change from baseline in monthly menstrual blood loss (MBL) to menstrual Cycle 3 | Baseline and end of menses Cycle 3 (approximately 12 weeks)
  MBL will be measured from blood collected from menstrual cycle by-products and recovered by alkaline hematin method during each menstrual cycle
Number of subjects with adverse events (AE) | Up to 3 months
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product; safety and tolerability as assessed by incidence of adverse events

SECONDARY OUTCOMES:
Change from baseline in monthly menstrual blood loss (MBL) at menstrual Cycle 1, 2, and 3 | Baseline, and end of menses Cycle 1, 2, and 3 (approximately 12 weeks)
  MBL will be measured from blood collected from menstrual cycle by-products
Average daily dysmenorrhea score from Day -1 to Day 2 in each cycle | Up to 3 months
  Average daily dysmenorrhea score from Day -1 to Day 2 of menses

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (13):
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Mandeville, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Lawrenceville, New Jersey
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Englewood, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas